CLINICAL TRIAL: NCT03311100
Title: Study of the Immunological Profile of Archival Formalin-fixed Paraffin-embedded Solid Tumors Sample
Brief Title: Immunological Profile of Solid Tumors Sample
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: Innate Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-53; 2017-A00778-45 (Registry Identifier: ID RCB)
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Solid Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Samples in formalin-fixed paraffin-embedded material block
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Lung cancer
  Interventions: Other: immunohistochemistry assay
- Central Nervous System Cancers
  Interventions: Other: immunohistochemistry assay
- Head and Neck and upper aero-digestive tract cancers
  Interventions: Other: immunohistochemistry assay
- Skin cancers
  Interventions: Other: immunohistochemistry assay
- Sarcomas
  Interventions: Other: immunohistochemistry assay
- Urothelial cancer
  Interventions: Other: immunohistochemistry assay
- Hepatocarcinoma
  Interventions: Other: immunohistochemistry assay

INTERVENTIONS:
Other: immunohistochemistry assay — biomarkers expression

SUMMARY:
It has become clear in the recent year that the nature of the immune cells infiltrate within a tumor was essential in the control of the tumor growth. This so-called immune contexture does vary between cancer types and in response to treatments. In this context, this trial is a non-interventional, mono-centric in patients with solid tumors. Samples in paraffin-embedded material block of biopsies or surgical pieces (either primitive tumor or metastases) will be analysed. For each sample, clinically relevant data associated with treated cancer and needed for characterization of tumor microenvironment will be documented.

This trial is, through accessing to well documented selected archival tumor materials, to validate selected biomarker for early phase trial.

ELIGIBILITY:
Inclusion Criteria:

* Sample must have had a valid written informed consent for available archival tumor samples for scientific purposes.
* Sample from patients with histologically documented cancer in target population.

Exclusion Criteria:

* Samples from subject unwilling to give their informed consent;
* Unusable sample or biologically deteriorated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid cancer
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Estimated)
Dates: Start 2017-04-06 (Actual); Primary Completion 2019-04-06 (Estimated); Study Completion 2020-04-06 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemistry scores | 24 months
  The immunohistochemistry scores is evaluated with the score of the percentage of stained cells.
  Scale of the score of the percentage of stained cells, From 0 to 4, 0 : no stained cell (absence)
  1. : < 10 % stained cell (minimal)
  2. : 10 to 50 % (mild)
  3. : 51 to 79 % (moderate)
  4. : = or > 80 % (marked)
Immunohistochemistry scores | 24 months
  The immunohistochemistry scores is evaluated with the score of the staining intensity.
  Staining Intensity: from 0 to 3 0 : no staining (absence)
  1. : low staining
  2. : middle staining
  3. : high staining

CONTACTS AND LOCATIONS:
Overall Officials: ARNAUD Jean-Olivier, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France